CLINICAL TRIAL: NCT05388812
Title: Individual Placement and Support for Veterans With Opioid Use Disorder: A Mixed Methods Study
Brief Title: Together in Recovery With Veterans Through Employment
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D3656-R
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Veterans With Opioid Use Disorder
Keywords: Veteran; opioid use disorder; employment; social support; mental health
MeSH Terms: conditions — Opioid-Related Disorders; Psychological Well-Being | interventions — Therapeutics; Palliative Care

STUDY DESIGN:
Intervention Model Description: eligible and consenting participants will be randomized to either individual placement and support (IPS) or treatment as usual vocational rehabilitation (TAU-VR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual Placement and Support (Experimental): The IPS model involves the following important domains: competitive employment, eligibility based on client choice of employment, integration of IPS and treatment team personalized counseling, rapid job search, systematic job development, and time-unlimited and individualized support.
  Interventions: Other: Individual Placement and Support (IPS)
- Treatment As Usual Vocational Rehabilitation (TAU-VR) (Active Comparator): TAU-VR Services may include 1) Compensated Work Therapy-Transitional Work (CWT-TW) assignment in a set-aside, minimum-wage, short-term job, typically in the VA setting (approximately 50% of the Veterans randomized to TW in past studies conducted by the investigators actually engaged in TW assignment) or 2) CWT-Community-Based Employment Services (CWT-CBES) which involves a community job search, placement in a competitive job, with limited follow-along support that typically ends after the Veteran is working in his/her first job
  Interventions: Other: Treatment As Usual Vocational Rehabilitation (TAU-VR)

INTERVENTIONS:
Other: Treatment As Usual Vocational Rehabilitation (TAU-VR) — TAU-VR Services may include 1) Compensated Work Therapy-Transitional Work (CWT-TW) assignment in a set-aside, minimum-wage, short-term job, typically in the VA setting (approximately 50% of the Veterans randomized to TW in past studies conducted by the investigators actually engaged in TW assignment) or 2) CWT-Community-Based Employment Services (CWT-CBES) which involves a community job search, placement in a competitive job, with limited follow-along support that typically ends after the Veteran is working in his/her first job
  Arms: Treatment As Usual Vocational Rehabilitation (TAU-VR)
Other: Individual Placement and Support (IPS) — The IPS model involves the following important domains: competitive employment, eligibility based on client choice of employment, integration of IPS and treatment team personalized counseling, rapid job search, systematic job development, and time-unlimited and individualized support.
  Arms: Individual Placement and Support

SUMMARY:
The purpose of this study is to help Veterans who have opioid use problems with gaining and maintaining meaningful employment. The investigators also want to know employment helps with other aspects of the Veteran's life including starting and staying on necessary medications, mental health needs, and feeling a part of society.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the employment outcomes of Individual Placement and Support (IPS) compared to Treatment-as-Usual Vocational Rehabilitation (TAU-VR) in 120 Veterans who are recovering from opioid use disorder (OUD) over 15 months. Specifically, the investigators will see which treatment yields more weeks worked in a competitive job with the hypothesis that IPS will result in better outcomes than TAU-VR. The investigators will interview Veterans in both IPS and TAU-VR groups to investigate the contextual barriers and facilitators of implementing vocational services among Veterans with OUD with the aim to provide solutions and leverage facilitators of success as the VHA expands supported employment services to a new priority population. Investigators will evaluate the impact of vocational services on adherence to prescribed treatment and OUD relapse rates. This study is especially timely given the societal impact of the COVID-19 pandemic on employment and occupational functioning.

ELIGIBILITY:
Inclusion Criteria:

* age 19* (<19 year of age in the state of AL is defined minor)
* DSM-5 Axis I diagnosis of OUD
* currently unemployed or underemployed, defined as working <20hrs/week in a meaningful competitive job for a wage, salary, or commission
* expression of interest in competitive employment; and willing and able to give informed consent

Exclusion Criteria:

* current diagnosis of psychotic disorders since these Veterans already can receive IPS in usual care at TVAMC and BVAMC
* diagnosis of dementia (evidenced in the medical record)
* presence of current severe and unstable medical condition or terminal illness, that would contraindicate study participation or expose them to an undue risk
* unlikely that participant can complete the study

  * e.g., expected deployment, incarceration, long-term hospitalization, or relocation from the vicinity
* active suicidal or homicidal ideation making it unsafe for Veteran to be included
* current participation in another vocational interventional trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
number of weeks worked | 15 months
  A "week worked" is defined as working either part time or full time in a competitive job during a Sunday to Saturday 7-day window. Competitive employment is defined as a job that pays at least minimum wage or is based on salary or commission, is based in a setting alongside others without disabilities, and is not reserved for people with disabilities

SECONDARY OUTCOMES:
Quality of Life | 15 months
  Veteran quality of life will be measures by a 16-item self-report quality of life scale by Burckhardt and Anderson. Scores range from 16 to 112. Higher numbers mean better quality of life. According to the authors, the average score of a healthy adult is 90. Therefore anything above 90 should be considered good.
social support | 15 months
  the Veterans perceived social support will be measured by the 37-item self-report community assessment inventory by Salari et al. There are four domains: household, (six items), family (10 items), friends 8 items), and community (13 items). scores can be calculated for each domain or on a total scale. for the total scale scores range from. Higher numbers mean higher perceived social support. No specific guidance on what is considered good or poor social support.
Depression | 15 months
  the Veterans depressive symptoms will be measured by the 9-item self-report Patient Health Questionnaire-9 by Pfitzer. Scores range from 1-27. Higher numbers mean more depressive symptoms. 1-4 is considered minimal depression; 5-9 is considered mild depression; 10-14 is considered moderate depression; 15-19 is considered moderately severe depression; and 20-27 is considered severe depression.
Anxiety | 15 months
  the Veterans anxiety will be measured by the 7-item self-report Generalized Anxiety Disorder-7 questionnaire by Spitzer et al. Scores range from zero to 21. Higher numbers mean more anxiety. zero to 4 is considered minimal anxiety; 5-9 is considered mild anxiety; 10-14 is considered moderate anxiety, and 15-21 is considered severe anxiety.
Resilience | 15 months
  the Veterans resilience will be measured by the 6-item self-report Brief Resilience Scale questionnaire by Smith et al. scores range from zero to 30 and then averaged by the number of questions answered. Therefore final scores averages range rom zero to 5. Higher mean scores reflect more resilience. The authors of the questionnaire do not provide any guidance on what is considered high, medium, or low resilience.

OTHER OUTCOMES:
suicide risk | 15-months
  the Veterans suicide risk will be measured by the self-report Columbia Suicide Severity Rating Scale (C-SSRS). The C-SSRS has three subscales' suicidal ideation, intensity of ideation, and suicidal behavior. Suicidal ideation subscale has 5 questions (yes/no). Intensity is rated 1-5 with most severe at 5; frequency is rated zero to 4 (0=not applicable; 1=only one time; 2=a few time; 3=a lot; 4=all the time). Suicidal behavior subscale is divided into actual attempt, interrupted attempt, aborted attempt or self-interrupted attempt, preparatory acts or behavior, and suicide. This is not a scored measure. This is a safety measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mercy N Mumba, RN, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama

IPD SHARING:
Plan to Share IPD: No